CLINICAL TRIAL: NCT03254849
Title: Effects on Blood Pressure and Central Sympathetic Nerve Traffic by SGLT2-inhibition With Empagliflozin Compared to Hydrochlorothiazide in Patients With Type 2 Diabetes Mellitus
Brief Title: Empagliflozin and Sympathetic Nerve Traffic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00/0764-Empa2
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- empagliflozin 25 mg (Experimental): Each patient will take 2 tablets each day to ensure double-blind Treatment. Arm 1: 25 mg/d empagliflozin + hydrochlorothiazide placebo
  Interventions: Drug: Empagliflozin
- hydrochlorothiazide 25 mg (Experimental): Each patient will take 2 tablets each day to ensure double-blind Treatment. Arm 2: 25 mg/d hydrochlorothiazide + empagliflozin placebo
  Interventions: Drug: Hydrochlorothiazide 25 mg

INTERVENTIONS:
Drug: Empagliflozin — 1 tablet
  Other Names: Jardiance
  Arms: empagliflozin 25 mg
Drug: Hydrochlorothiazide 25 mg — 1 tablet
  Other Names: HCT
  Arms: hydrochlorothiazide 25 mg

SUMMARY:
In this study the effects of the Inhibition of the Sodium-Glucose Linked Transporter 2 in the kidney with empagliflozin compared to hydrochlorothiazide on blood pressure and on central sympathic nervous activity will be examined.

DETAILED DESCRIPTION:
The drug empagliflozin is a selective oral inhibitor of the sodium-glucose co-transporter 2 (SGLT-2) in the kidney.On the market empagliflozin is approved for the treatment of type 2 Diabetes. The mechanism of action can be described as follows: SGLT-2 is responsible for 90% of the reabsorption of Glucose in the kidney. If this Transport System is inhibited the secretion of glucose via the urine is increased. Therefore the blood glucose concentration will be lowered.

It has been noted that the SGLT-2 drugs are lowering the blood pressure as well, but the specific characteristics of the durg leading to this effect have not been examined in adequate clinical trial up to now.

To evaluate the central sympathic nervous activity a microneurography will be performed in this study; this examination will provide Information if empagliflozin dose decrease the sympathic nervous activity. If this is the case new effects of empagliflozin have to be discussed, Otherwise it can be assumed that the blood pressure decrease is a result of an increase of urine volume. In this case the sympathic activity should be increased.

This study will be performed in parallel groups who will receive a double-blind, randomised treatment, either empagliflozin or hydrochlorothiazide. The hypothesis that empagliflozin - in contrast to hydrochlorthiazide - does not increase the sympathic nervous activity in obese, hypertensive subjects with type 2 Diabetes treated with metformin will be tested.

ELIGIBILITY:
Inclusion Criteria:

* women and men >= 50 and <= 80 years of age
* type 2 diabetes mellitus for >=2 years
* only metformin monotherapy is allowed; metformin dose must have been stable for >=12 weeks

Exclusion Criteria:

* previous empagliflozin treatment within the last 3 months
* heart failure NYHA II - IV
* subjects who have received any investigational medicinal product or have used any investigational medical device within 30 days prior to the screening visit, or who are actively participating in any investigational medicinal product or medical device trial, or who are scheduled for any such trial during the course of the trial.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Blood Pressure reduction | 6 weeks
  Blood pressure reduction with empagliflozin treatment is associated with lesser increase in sympathetic nerve traffic when compared to Hydrochlorothiazide treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany